CLINICAL TRIAL: NCT06294106
Title: Electroencephalogram (EEG) Personalized Transcranial Magnetic Stimulation (eTMS) for Post-Traumatic Stress Disorder (PTSD)
Brief Title: eTMS for Veterans and First Responders With PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Wave Neuroscience (Industry)
Responsible Party: Principal Investigator, Wynn Legon, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 24-212
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: 10 participants will receive eTMS treatment 10 participants will receive sham eTMS treatment
Who Masked: Participant, Investigator
Masking Description: eTMS coil will have an 'active' and 'sham' side and the application will look identical to the participant. The technician will not know which side of the coil is which and will additionally be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- eTMS (Experimental): The active side of a TMS coil will be used to administer eTMS application.
  Interventions: Device: Electroencephalogram personalized Transcranial Magnetic Stimulation (eTMS)
- eTMS sham (Sham Comparator): The sham side of a TMS coil will be used to administer a sham dosage of eTMS application.
  Interventions: Device: Electroencephalogram personalized Transcranial Magnetic Stimulation (eTMS)

INTERVENTIONS:
Device: Electroencephalogram personalized Transcranial Magnetic Stimulation (eTMS) — EEG is utilized to determine a personalized frequency to then apply TMS to the frontal lobe.

SUMMARY:
A battery of physiological and behavioral data will be collected before and after application of eTMS. Participants will be veterans or first responders diagnosed with PTSD. Study will be a double-blind, sham-controlled, parallel group, randomized clinical trial.

DETAILED DESCRIPTION:
Veterans and first responders diagnosed with PTSD will be studied to evaluate safety and efficacy of an EEG personalized TMS paradigm. All participants will undergo 2 days of extensive testing prior to eTMS application and 2 days of testing after. Testing will include MRI, OPM, EEG, behavioral tasks, questionnaires, and an EEG sleep study.

ELIGIBILITY:
Inclusion Criteria:

* Veteran or first responder
* diagnosed with post-traumatic stress disorder with PCL-5 cutoff of 31 or above

Exclusion Criteria:

* Claustrophobia
* Contraindications to MRI
* Pregnant
* Uncontrolled medical, psychological, or neurological conditions
* Unable to calculate EEG alpha frequency
* History of ECT or rTMS
* History of intracranial lesion or increased intracranial pressure
* History of stroke
* History of other neurologic conditions
* Family history of epilepsy
* Personal history of epilepsy
* certain medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Up to 7 weeks
  Adverse event reports (or lack-of) will determine device safety
Report of Symptoms | Up to 7 weeks
  Symptom questionnaire to be completed before and after all study procedures to determine feasibility in this patient population. Various symptoms will be rated on a likert scale from absent to severe.

SECONDARY OUTCOMES:
PCL-5 | Up to 7 weeks
  Completion of the PTSD symptom questionnaire. Scores range from 0-80, with a PTSD cutoff score of 31.
fMRI | 1 session 1 week pre treatment and 1 session 1 week post treatment
  Functional MRI signals including BOLD signals collected at rest and during basic tasks to assess neuropathways of activation
OPM | 1 session 1 week pre treatment and 1 session 1 week post treatment
  Optically Pumped Magnetometry signals collected at rest and during basic tasks to assess neuropathways of activation
EEG | Up to 7 sessions collected over 7 weeks.
  Electroencephalography recordings at rest and during a stress task. Specifically analyzing the P300.

CONTACTS AND LOCATIONS:
Overall Officials: Wynn Legon, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Fralin Biomedical Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No